CLINICAL TRIAL: NCT07359170
Title: Impact of Elective Versus Emergency Cesarean Delivery on Early Postpartum Depression: a Retrospective Study
Brief Title: Delivery Mode Impact on Postoperative Depression
Status: Not yet recruiting | Type: Observational
Sponsor: Jingping Wang, MD, Ph.D. (Other)
Responsible Party: Sponsor-Investigator, Jingping Wang, MD, Ph.D., Associate Professor Staff Anesthesiologist & Pain Physician, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Other Study IDs: 2025P002461
Record Dates: First submitted 2026-01-14; First posted 2026-01-22 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Postoperative Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (3):
- elective cesarean: patients who undergone elective cesarean
- urgent cesarean: patients undergone urgent cesarean
- vaginal delivery: patients who delivered by vaginal pass

SUMMARY:
The goal of this observational retrospective cohort study is to examine the association between mode of delivery and early postpartum depressive symptoms in adult women who delivered at Massachusetts General Hospital. Specifically, the study evaluates whether the urgency of cesarean delivery (elective versus emergency) is associated with differences in Edinburgh Postnatal Depression Scale (EPDS) scores at 6-8 weeks postpartum, compared with elective cesarean delivery and vaginal delivery. The EPDS is a validated 10-item self-report questionnaire with scores ranging from 0 to 30, where higher scores indicate more severe depressive symptoms.

The primary questions are whether EPDS scores differ among women undergoing emergency cesarean delivery, elective cesarean delivery, and vaginal delivery, and whether perioperative and obstetric factors are associated with postpartum depressive symptoms.

This study involves retrospective analysis of de-identified electronic health record data. Participants will not undergo any study-specific interventions.

ELIGIBILITY:
Inclusion Criteria:

Underwent cesarean delivery (elective or emergency) or vaginal delivery during the study period

Age 18 years or older

Completed at least one Edinburgh Postnatal Depression Scale (EPDS) assessment at 6-8 weeks postpartum

Have complete perioperative data available

Exclusion Criteria:

Missing 6-8 week postpartum EPDS scores

Pregnancy with fetal demise, severe obstetric complications, or atypical maternal conditions

History of severe psychiatric disorders (e.g., schizophrenia, bipolar disorder), when identifiable

Incomplete perioperative medical records

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients (≥18 years old) who underwent cesarean delivery or vaginal delivery
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Edinburgh Postnatal Depression Scale (EPDS) scores, a 10-item self-reported screening tool for postpartum depression (range: 0-30, with higher scores indicating more severe depressive symptoms) | 6-8 weeks postpartum

SECONDARY OUTCOMES:
Prevalence of postpartum depression | 6-8weeks
  Prevalence of postpartum depression (EPDS ≥ threshold) across delivery groups.